CLINICAL TRIAL: NCT00452595
Title: A 12-Month Open-Label Evaluation of the Long-Term Safety of DVS-233 SR in Outpatients With Major Depressive Disorder
Brief Title: Study Evaluating DVS-233 for Treatment of Outpatients With Major Depressive Disorder
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 3151A1-318
Record Dates: First submitted 2007-03-23; First posted 2007-03-27 (Estimated); Last update posted 2007-03-27 (Estimated); Status verified 2007-03

CONDITIONS: Major Depressive Disorder
MeSH Terms: conditions — Depressive Disorder, Major

INTERVENTIONS:
Drug: DVS-233 SR (desvenlafaxine sustained release )

SUMMARY:
To evaluate the long-term safety of desvenlafaxine sustained release (DVS-233SR) during open-label treatment of outpatients with major depressive disorder (MDD).

ELIGIBILITY:
Inclusion Criteria:

* Outpatients.
* Men and women aged 18 to 75 years.
* Women of childbearing potential must have a negative serum pregnancy test result at screening. Sexually active individuals participating in this study must use a medically acceptable form of contraception during the study and for at least 15 days after the last dose of test article.
* Subjects must have a primary diagnosis of MDD based on the criteria in the Diagnostic and Statistical Manual of Mental Disorders, 4th edition (DSM-IV), single or recurrent episode, without psychotic features, on study day 1. If other allowable psychiatric diagnoses are present, MDD must be the predominant psychiatric disorder present. (See Exclusion Criterion 6 for psychiatric diagnoses that are not allowable.)
* Depressive symptoms for at least 30 days before the screening visit.
* Subjects who have symptoms of depression judged by the investigator to require long-term treatment (i.e., 6 months or longer) with an antidepressant drug.

Other inclusion applies.

Exclusion Criteria:

* Treatment with DVS-233 SR at any time in the past.
* Treatment with venlafaxine (immediate release [IR] or extended release [ER]) within 90 days of study day 1.
* Known hypersensitivity to venlafaxine (IR or ER).
* Significant risk of suicide based on clinical judgment, including common suicidal thoughts, and suicide being considered as a possible solution, even without specific plans or intention.
* Women who are pregnant, breastfeeding, or planning to become pregnant during the study.
* Current (within 12 months of baseline) psychoactive substance abuse or dependence (including alcohol), manic episode, posttraumatic stress disorder, obsessive-compulsive disorder, or a lifetime diagnosis of bipolar or psychotic disorder as assessed by the modified Mini International Neuropsychiatric Interview (MINI). Current (within 12 months of baseline) generalized anxiety disorder, panic disorder, or social anxiety disorder as assessed by the modified MINI and considered by the investigator to be primary, causing a higher degree of distress or impairment than MDD. Presence (within 12 months of baseline) of a clinically important personality disorder (such as antisocial, schizotypal, histrionic, borderline, narcissistic).
* Depression associated with the presence of an organic mental disorder due to a general medical condition or a neurologic disorder.
* History of a seizure disorder other than a single childhood febrile seizure.

Other exclusion applies.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2004-01; Study Completion 2005-05

PRIMARY OUTCOMES:
HAM-D17

SECONDARY OUTCOMES:
MADRS, CGI-S, CGI-I, Covi Anxiety Scale, SDS, VAS-PI, and WHO-5

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Wyeth is now a wholly owned subsidiary of Pfizer